CLINICAL TRIAL: NCT06193993
Title: Low-dose 500 mg Abiraterone Acetate in Metastatic Castration-resistant Prostate Cancer (mCRPC) and Metastatic Hormone-sensitive Prostate Cancer (mHSPC) Patients: a Phase I Proof-of-concept Clinical Study
Brief Title: Effect of Low-dose 500 mg Abiraterone Acetate in Treatment of Metastatic Prostate Cancer Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NUH-DSRB-2020/00258
Record Dates: First submitted 2023-12-05; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer; Metastatic Cancer; Hormone Sensitive Prostate Cancer; Castration-resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abiraterone Acetate (Experimental): 500 mg dose of Abiraterone Acetate plus prednisolone
  Interventions: Drug: Abiraterone Acetate

INTERVENTIONS:
Drug: Abiraterone Acetate — Upon successful registration, patients would be initiated on 500 mg once daily (two 250 mg tablets), plus prednisolone 5 mg twice daily orally for mCRPC and 5mg once daily orally for mHSPC.

SUMMARY:
This will be an open label, Phase I study to assess the efficacy of a reduced 500 mg dose of abiraterone acetate in patients with metastatic prostate cancer. Eligible metastatic hormone-sensitive prostate cancer (mHSPC) and metastatic castration-resistant prostate cancer (mCRPC) patients newly initiated on abiraterone acetate treatment will be recruited to receive a reduced 500 mg dose of abiraterone acetate plus prednisolone. The study treatment duration will span 12 weeks, after which patients being administered the reduced dose will be reverted to the standard 1000 mg dosing. Follow-up for mCRPC and mHSPC patients will last for 18 and 36 months respectively. The main question the study aims to answer is whether dose reduction of abiraterone acetate to 500 mg would achieve antitumor activity in mCRPC and mHPSC patients comparable to standard of care.

DETAILED DESCRIPTION:
Primary Objectives:

As a preliminary Phase I trial, the primary objective of the study would be to evaluate the percentage change in prostate specific antigen (PSA) from baseline to 12 weeks.

Secondary Objectives:

1. determine the proportion of patients achieving PSA response (≥ 50% reduction in PSA after 12 weeks of therapy).
2. evaluate the pharmacokinetics associated with the 500 mg dose of abiraterone acetate.
3. investigate the correlation between plasma exposure of abiraterone and CP-I or CP-III in order to support their utility as a biomarker of OATP1B1/1B3 function.
4. assess the pharmacodynamic effects of the reduced 500 mg dose on the maximal percentage change in serum androgens (dehydroepiandrosterone (DHEA), dehydroepiandrosterone-sulfate (DHEA-S), testosterone, androstenedione) from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma prostate
2. Age >21 years
3. Diagnosis of metastatic castration-resistant prostate cancer (mCRPC) (chemotherapy naïve and chemotherapy pre-treated patients) or metastatic hormone-sensitive prostate cancer (mHSPC)
4. For mCRPC patients, evidence of castration resistance is defined as disease progression despite a testosterone level <50ng/dL (or surgical castration)
5. Progressive disease was defined as either

   1. PSA progression according to Prostate Cancer Working Group (PCWG2) criteria15: PSA evidence for progressive prostate cancer consists of a minimum PSA level of at least 2 ng/ml, which has subsequently risen on at least 2 successive occasions, at least 1 week apart
   2. Radiographic progression according to RECIST 1.1 guidelines or
   3. 2 or more new lesions on bone scan
6. Newly initiated on abiraterone acetate therapy
7. Eastern Cooperative Oncology Group (ECOG) performance status grade of 0, 1 or 2.
8. Adequate hematologic, hepatic, and renal function would include:

   * hemoglobin ≥9.0 g/dL independent of transfusions
   * neutrophils ≥1.5 x 109/L
   * platelets ≥100 x 109/L
   * total bilirubin ≤1.5× upper limit of normal (ULN) [except for subjects with documented Gilbert's disease in which case total bilirubin not to exceed 10× ULN]
   * alanine (ALT) and aspartate (AST) aminotransferase ≤2.5X ULN
   * serum creatinine <1.5× ULN or calculated creatinine clearance ≥30 mL/min
   * serum potassium ≥3.5 mmol/L
9. Ability to provide informed consent

Exclusion Criteria:

1. Patients with prior use of enzalutamide or other potent androgen pathway targeted therapies
2. Concurrent therapy with strong inhibitors or inducers of CYP3A4 due to concerning possible drug-drug interactions with abiraterone.
3. Concurrent therapy with strong inhibitors or inducers of OATP transporters (e.g., rifampicin, cyclosporine) due to concerning possible effects on CP-I and CP-III.
4. New York Heart Association (NYHA) class II, NYHA class III, or IV congestive heart failure (any symptomatic heart failure)
5. Uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic BP ≥95 mmHg). Subjects with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
6. Patients who do not voluntarily consent to participate in the study

Ages: 21 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with greater than or equal to 50 percent decrease in Prostate Specific Antigen (PSA) levels | Baseline up to Week 12

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of 500 mg dose of Abiraterone Acetate | Pre-dose and 0.5, 1, 2, 3, 4 and 6 hours post-dose on Visit 1 (Week 2 from start of treatment)
Time to Reach the Maximum Plasma Concentration (Tmax) of 500 mg dose of Abiraterone Acetate | Pre-dose and 0.5, 1, 2, 3, 4 and 6 hours post-dose on Visit 1 (Week 2 from start of treatment)
Area under the plasma concentration time curve from time 0 to 6 hours (AUC0-6h) of 500 mg dose of Abiraterone Acetate | Pre-dose and 0.5, 1, 2, 3, 4 and 6 hours post-dose on Visit 1 (Week 2 from start of treatment)
Area under the plasma concentration time curve from time 0 to infinity time (AUC0-inf) of 500 mg dose of Abiraterone Acetate | Pre-dose and 0.5, 1, 2, 3, 4 and 6 hours post-dose on Visit 1 (Week 2 from start of treatment). On Visits 2 (Week 4), 3 (Week 8) and 4 (Week 12) pre-dose
Volume of distribution (Vd) of 500 mg dose of Abiraterone Acetate | Pre-dose and 0.5, 1, 2, 3, 4 and 6 hours post-dose on Visit 1 (Week 2 from start of treatment). On Visits 2 (Week 4), 3 (Week 8) and 4 (Week 12) pre-dose
Apparent oral clearance (CL/F) of 500 mg dose of Abiraterone Acetate | Pre-dose and 0.5, 1, 2, 3, 4 and 6 hours post-dose on Visit 1 (Week 2 from start of treatment). On Visits 2 (Week 4), 3 (Week 8) and 4 (Week 12) pre-dose
Trough plasma concentrations at steady state (Ctrough) of 500 mg dose of Abiraterone Acetate | Baseline up to Week 12
Plasma concentrations of testosterone | Baseline up to Week 12
Plasma concentrations of androstenedione | Baseline up to Week 12
Plasma concentrations of dehydroepiandrosterone-sulfate (DHEA-S) | Baseline up to Week 12
Plasma concentrations of cortisol | Baseline up to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Chiong, MBBS, PhD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No